CLINICAL TRIAL: NCT04581226
Title: 'Correlation Between Lung Ultrasound Findings and Clinical Consequences of High Intraoperative Inspired Oxygen Fraction During Elective Surgery in Mechanically Ventilated Children''
Brief Title: LUS and Consequences of High FiO2 in Children
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Professor of anesthesia and intensive care, Assiut University
Other Study IDs: 17101201
Record Dates: First submitted 2020-09-20; First posted 2020-10-09 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Perioperative/Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lung ultrasound: Sonographic assessments including the lung consolidation score, B-line score and Lung aeration score will be recorded 1min. after intubation, at end of surgery and 2h postoperatively.
  Interventions: Diagnostic Test: Lung ultrasound

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — All children will be studied in the supine position. LUS will be performed with the portable device MicroMax (Sonosite, Bothell, Washington, USA) using a linear probe of 6 to 12 MHz. All ultrasound scans will be performed by the same anesthetist, who has experience of more than 30 lung ultrasound scans in pediatric patients. Each hemithorax will be divided into six regions, using three longitudinal lines (parasternal, anterior and posterior axillary) and two axial lines (one above the diaphragm and the other 1 cm above the nipples)
  Other Names: Lung Sonar

SUMMARY:
The purpose of this study is

1. to evaluate effect of high FiO2 on the development of intraoperative atelectasis in mechanically ventilated children using LUS.
2. to investigate the correlation between lung consolidation score and patient clinical variables including pulmonary mechanics, Sao2%, ABG, and perioperative respiratory complications.

DETAILED DESCRIPTION:
The WHO and United States centers for disease control and prevention (CDC) recently recommended the administration of 80% inspired oxygen fraction (Fio2) during and immediately after surgery performed with general anesthesia and endotracheal intubation.

The recommendation was based on some data suggesting that intra-operative high Fio2 reduces incidence of surgical site infections.

The dilemma of applying high or low perioperative FiO2 arises in daily practice of pediatric anesthesia because children are at increased risk of developing hypoxemia due to their physiological characteristics including smaller functional residual capacity and increased metabolic requirement compared with adult.

However, considering that atelectasis occurs in most pediatric patients undergoing general anesthesia, it is important to titrate perioperative level of FiO2 to minimize the risk of developing atelectasis and hypoxemia.

The use of FiO2 80% at induction and emergence, whilst limiting FiO2 to 35% during maintenance of anesthesia, may prevent the occurrence of atelectasis and ensure sufficient oxygenation.

Conversely, the use of FiO2 100% at induction and emergence, which is reduced to FiO2 80% during maintenance of anesthesia, may increase the margin of safety to avoid hypoxemia.

In children, the pulmonary consequences of using high FiO2 during general anesthesia have not been fully characterized over the early perioperative period. LUS has shown reliable sensitivity and specificity for diagnosis of anesthesia-induced atelectasis in children [7]. It can identify children needing a recruitment maneuver to re expand their lung and help optimize ventilator treatment during anesthesia.

Our hypothesis is that clinical data are necessary to validate the lung sonographic findings of atelectasis and negative consequences of administrating high perioperative oxygen concentration.

ELIGIBILITY:
Inclusion criteria:

* Age of 1-6 years.
* ASA physical status (I-II).
* Endotracheal intubation and mechanical ventilation.
* Elective non-abdominal and non-thoracic surgery
* lasting for more than 2 hours.

Exclusion criteria:

* ASA classification more than II
* Thoracic or abdominal surgery.
* pre-existing lung disease.
* Pre-operative chest infection or abdominal chest US finding. Any thoracic deformity Patients with cardiac, liver or kidney disease.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Age of 1-6 years.
  * ASA physical status (I-II).
  * Endotracheal intubation and mechanical ventilation.
  * Elective non-abdominal and non-thoracic surgery
  * lasting for more than 2 hours.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
LUS-consolidation Score | It will be recorded intraoperative to 2hours postoperative.
  The lung ultrasound consolidation score that is divided into four grades and scored between 0 and 3: (0) no consolidation; (1) minimal juxta-pleural consolidation; (2) small-sized consolidation; and (3) large-sized consolidation. Anesthesia-induced atelectasis will be defined to be significant if any region had a consolidation score of ≥ 2.

SECONDARY OUTCOMES:
LUS-B-line Score | It will be recorded intraoperative to 2hours postoperative.
  Lung ultrasound B-Line score. The degree of B-lines will be assessed by the ''B-lines score'' that is divided into four grades and scored between 0 and 3: (0) fewer than three isolated B-lines; (1) multiple well-defined B-lines; (2) multiple coalescent B-lines; and (3) white lung,

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Professor of anesthesia and intensive care.
Locations (2):
- Egypt (2):
  - Assiut university Pediatric hospital, Asyut, Assiut Governorate
  - Hala Abdel-Ghaffar, Asyut, Asyut Governorate

IPD SHARING:
Plan to Share IPD: No